CLINICAL TRIAL: NCT04905472
Title: Vestibular Implants Tested in Human Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic during the 1year of grant funding (2019-2020), no new patients were implanted with the vestibular prosthetic device and enrolled in this study at the University of Geneva study site.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Ohio State University (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Richard Lewis, Associate Professor, Otolaryngology and Neurology; Director, Jenks Vestibular Laboratory, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019A008661
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Vestibular Disorder; Vestibular Ataxia; Vestibular Loss, Bilateral
Keywords: eye movements; perception; vestibular; dizziness; sensory integration; prosthesis
MeSH Terms: conditions — Vestibular Diseases; Bilateral Vestibulopathy; Dizziness | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibular & Cochlear Implant Patients (Experimental): * scheduled for CI surgery because of deafness
  * a minimum of five year history of documented absence of auditory and vestibular function, based on review of their audiograms and vestibular tests.
  * Specific vestibular criteria are: peak ice water caloric response of less than 3 deg/s for each ear; yaw VOR time constant < 3.0 sec and gain < 0.25; and reduced head impulse gain (<0.25) for all canal planes.
  * Specific audiographic criteria: 80dB or greater sensorineural hearing loss in both ears
  Interventions: Device: Vestibular prosthesis/implant; Device: Vestibular Implant Stimulation

INTERVENTIONS:
Device: Vestibular prosthesis/implant — The intervention is a vestibular prosthesis which our collaborators at the University of Geneva are implanting into the inner ear in deaf patients without vestibular function who are receiving a cochlear implant. The vestibular implant (VI) has three rate sensors and senses angular head velocity in three dimensions and provides this information to the brain by stimulation the afferent nerves innervating the three semicircular canals. Our goal is to use the VI to better understand how the brain processes this prosthetic information and uses it to generate meaningful behavioral responses including eye movements, postural control, and perception.
Device: Vestibular Implant Stimulation — VI subjects will be studied before the implant is activated (pre) and then after it is turned on (acute On); this will take about 2 hrs. Then they will have 8 hours of motion-modulated VI stimulation while they actively explore the hospital environment, after studies will be repeated (chronic On). Each set of outcome experiments will be performed twice, once with and once without low-levels of stochastic noise added to the VI stimulation provided for the 8-hour period. The noise amplitude is tailored to each patient to maximize stochastic resonance so extraction & integration of spatial signal provided by the VI will always be the first experiment, but the order of the subsequent outcome sessions (active/passive head rotations, tilt/translation motion discrimination and VOR behavioral changes & postural control) will be randomized. VI subjects will participate in 4 full-day sessions, each separated by at least a month.

SUMMARY:
The goal of this study is to improve the vestibular implant's ability to reduce the vestibular-dependent perceptual, postural, and visual symptoms that affect patients with severe peripheral vestibular damage. The long-term research plan is focused on exploring the three questions which must be answered to assess the clinical utility of a vestibular implant (VI) in vestibulopathic patients - i) how can information transfer from the VI sensors to the brain be optimized; ii) how does the three-dimensional angular velocity information provided by the VI interact in the brain with other sensorimotor (vision, otolith, efferent) signals; and iii) how effectively does the VI alleviate the behavioral deficits and subjective symptoms experienced by patients with severe vestibular damage. The current study will be used to focus on two key subsets of these questions. Over one year, the investigators will study approximately 5 patients who have severe bilateral vestibular damage and functioning VI's, which will focus on aim 1: how the angular velocity information sensed by the VI can be optimally transferred to the brain; and aim 2: how effectively the VI improves the clinical status of vestibulopathic patients when they receive acute and sub-acute (3 days) motion-modulated stimulation. In sum, the investigators aim to improve the efficacy of the VI in human subjects by developing new knowledge about how the brain processes motion cues provided by the VI and correlating this information with behavioral outcomes.

DETAILED DESCRIPTION:
Aim1: Optimizing information transfer from the VI to the brain: the investigators will study two approaches - altering the transfer function that relates the head's angular velocity to the electrical stimulation applied by the VI to the canal ampullary nerves; and utilizing the VI's unique capability to add noise to vestibular afferents. Regarding the former, the study team plans to initiate investigation of the principal components of the transfer function by testing the VI's capabilities when - the baseline resting stimulation rate is modified up or down; the temporal filtering (e.g., corner frequency of the high-pass filter) of the angular velocity signal recorded by the rate sensor is modified; the slope of the linear component of the hyperbolic tangent function that relates filtered head velocity to stimulation strength is altered; and different modes of stimulation modulation are used to encode head velocity (e.g, modifying the amplitude, the rate, or co-modulating the amplitude and rate of the current pulses). Regarding the use of noise, the investigators will test a given transfer function with different amplitudes of broad-band white electrical noise superimposed on the stimulation that encodes angular velocity, to determine if information transfer can be improved from the VI to the brain with low-level noise via stochastic resonance, as has been demonstrated in other sensory systems. To determine the efficacy of these approaches, the study team will measure the three basic vestibular-mediated behaviors (eye movements, posture, and perception). In particular we will focus on the amplitude and threshold of the angular vestibulo-ocular reflex (VOR), yaw-axis perceptual thresholds, and postural sway thresholds and amplitude, with the goal of defining the transfer function and noise level that minimizes thresholds (e.g., optimizes the signal-to-noise ratio) and maximizes the amplitude of the behavioral responses. One corollary of these studies is to examine if the different behavioral pathways are optimized with different stimulus parameters, as is suggested by the preliminary data.

Aim 2: Characterizing the effects of VI stimulation on clinical status: Vestibular-mediated behaviors are crucial to patient wellbeing and are degraded after severe vestibular damage. The investigators will initiate the assessment of the VI's clinical utility by quantifying the VOR, posture/gait, and perception using paradigms that isolate the VI's contributions to these behaviors (e.g., VOR during yaw-axis rotation) or paradigms that recapitulate normal activities such as self-generated walking, which require the brain to synthesize the angular velocity information provided by the VI with other sensorimotor cues. The investigators will study these vestibulopathic patients before the VI is activated ('pre'), one hour after activation ('acute,' which allows participants adequate time to adapt to the tonic VI stimulation), and then daily for three days while motion-modulated stimulation is provided by the VI during normal activities ('chronic'). The investigators will also have participants complete several questionnaires prior to stimulation and again in the acute and chronic stimulation states to quantify their subjective responses to VI stimulation. These will include questionnaires that characterize the severity of subjective dizziness and imbalance (Dizziness Handicap Inventory [DHI], Activities Specific Balance Confidence Scale [ABC]); oscillopsia (the Oscillopsia Functional Impact Scale); and a more general quality of life measurement (the Short Form-36 Health Survey). These questionnaires will be modified so they reflect current levels of symptomatology, since the study team will be capturing changes over a short time-frame. The investigators expect that behavior and symptoms will improve during the period of motion-modulated stimulation such that measurements and subjective reports in the 'chronic' stimulation state will be closer to normal than during the 'acute' or 'pre' stimulation states. More complex behaviors (e.g. balance while walking, ABC scores) are predicted to improve more slowly than behaviors that rely on isolated angular velocity cues (e.g., yaw axis VOR, oscillopsia scores). In sum, this study will provide a solid foundation to build upon for future research in which the investigators will further examine the clinical utility of the VI.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cochlear implant CI surgery because of deafness
* minimum of five year history of documented absence of auditory & vestibular function, based on review of their audiograms & vestibular tests
* Specific vestibular criteria are: peak ice water caloric response of less than 3 deg/s for each ear; yaw VOR time constant < 3.0 sec and gain < 0.25; and reduced head impulse gain (<0.25) for all canal planes.
* Specific audiographic criteria: 80dB or greater sensorineural hearing loss in both ears

Exclusion Criteria:

* pregnant
* not scheduled for cochlear implant/vestibular implant surgery
* unable to walk 50m
* other neurological disorder (other than migraine), otologic disease (other than presbycusis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in Postural Sway Thresholds | 3 days
  Changes in threshold for postural sway, measured using IMUs (inertial measurement unit) placed on the upper back, head, and torso, will be assessed before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following motion-modulated stimulation.
Changes in Postural Sway Amplitudes | 3 days
  Changes in amplitude in postural sway, measured using IMUs (inertial measurement unit) placed on the upper back, head, and torso, will be assessed before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following motion-modulated stimulation.
Changes in Gait dynamics | 3 days
  Changes in gait dynamics, measured using IMUs (inertial measurement unit) placed on the upper back, head, each ankle, and torso during various physical therapy walking tasks (Functional Gait Analysis), will be assessed before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following motion-modulated stimulation.
Changes in Vestibular Ocular Reflex (VOR) Amplitude | 3 days
  This reflex which moves the eyes in response to head movement and is driven by the sensors in the inner ear. Participants will walk in place while fixating on a cyclopean eye-centered near target (0.5m) and a far target (10m) for 60sec each. A lightweight infrared eye tracker with built in 6 degree of freedom IMU (eyeseecam) will be used to measure eye and head movements together. The amplitude or 'gain' (eye velocity divided by head velocity) is assessed before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation. Low gain is associated with impaired VOR.
Changes in Vestibular Ocular Reflex (VOR) Threshold | 3 days
  This reflex which moves the eyes in response to head movement and is driven by the sensors in the inner ear. Participants will wear a lightweight infrared eye tracker with built in 6 degree of freedom IMU (eyeseecam). Investigators will gently rotate the participant about the yaw-axis while measuring eye and head movements together. The velocity threshold for VOR is quantified before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following motion-modulated stimulation.
Changes in motion perception in yaw | 3 days
  Perception of head motion and orientation relative to gravity is measured by a continuous task during yaw rotation where the goal is to keep a light pointing in the direction of the start position/straight ahead. The task requires constant corrections because the light's orientation shifts randomly (based on integrated Brownian noise) and accelerates when a wheel is turned, resulting in overshooting errors. This method, a variant of the Critical Control Task used in humans, is an accurate way to capture perceived head motion. Motion perception during yaw-rotation will be assessed before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation.
Changes in motion perception orientation in roll | 3 days
  Perception of head motion and orientation relative to gravity is measured by a continuous subjective-visual-vertical (SVV) task where the subject uses a small steering wheel to keep a light bar orientated parallel to the perceived earth-vertical. The task requires constant corrections because the light bar's orientation shifts randomly (based on integrated Brownian noise) and accelerates when the wheel is turned, resulting in overshooting errors. This method, a variant of the Critical Control Task used in humans, is an accurate way to capture perceived head orientation. The 'perceived upright' is assessed before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation.
Changes in angular error during a navigation task | 3 days
  Participants will perform a path integration or 'complete the triangle' virtual reality task - angular error of responses is measured before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation. Greater angular error and variability of angular error is associated with worse visual-spatial memory.
changes in dizziness handicap index score | 3 days
  Participants will fill out the dizziness handicap index questionnaire before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation. It is scored 0 to 100 with high scores indicating greater subjective dizziness and disbalance.
changes in activities-specific balance confidence score | 3 days
  Participants will fill out the activities-specific balance confidence questionnaire before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation. It is scored from 0-100% with lower scores showing less confidence in balance and more subjective dizziness.
changes in oscillopsia functional impact scale score | 3 days
  Participants will fill out the oscillopsia functional impact scale before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation. It is scored from 0 to 215 in 5 point increments.
changes in reported quality of life | 3 days
  Quality of life will be assessed by participants filling out the short form-36 health survey (scored 0 to 100 points) before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation.
changes in cognitive impairment - visual-spatial function | 3 days
  Cognitive impairment will be assessed by participants completing a neuropsychological test battery with a focus on visual-spatial tasks before prosthetic stimulation, immediately after the prosthesis is activated, and daily for 3 days following 8hrs of motion-modulated stimulation. More errors and time to complete the tasks in the battery are associated with visual-spatial memory and function impairment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio
- Universite de Geneve Hospital (UNIGE), Geneva, Switzerland